CLINICAL TRIAL: NCT01014533
Title: This is a Study Exploring the Reasons Why People With Alcohol Dependence Have Sleep Disturbances, and Whether or Not a Study Medication, Gabapentin, vs. Placebo, Affects Those Sleep Patterns.
Brief Title: Pharmacotherapy and Mechanisms of Sleep Disturbance in Alcohol Dependence
Acronym: MA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Kirk Brower (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Dr. Kirk Brower, Professor of Psychiatry, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HUM00010947; 1R01AA016117-01A1 (NIH)
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Results first posted 2017-11-01 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-10

CONDITIONS: Alcohol Dependence; Insomnia
Keywords: Alcoholism; Alcohol dependence; Insomnia; Dim light melatonin onset; Gabapentin
MeSH Terms: conditions — Alcoholism; Sleep Initiation and Maintenance Disorders | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): After 3 nights in the UM sleep lab and randomization, this arm receives placebo for one week. They then return to the sleep lab for the same procedures.
  Interventions: Drug: Placebo dispensed to subject.
- Gabapentin (Active Comparator): After spending 3 baseline nights in the UM sleep lab, alcohol dependent subjects are randomized. This arm receives gabapentin . On nights 1 and 2 of medication, the dose is 600 mg by mouth 30 min before bedtime. On nights 3-10, the dose is 1200 mg by mouth 30 min before bedtime. On nights 8-10 of medication, subjects return to the UM sleep lab and complete 3 sleep nights with the same procedures. On night 11, the dose is reduced to 600 mg by mouth 30 min before bedtime, and then stopped.
  Interventions: Drug: Gabapentin dispensed to subject.

INTERVENTIONS:
Drug: Placebo dispensed to subject. — Placebo for 11 days, (one pill at bedtime on nights 1 and 2, 2 pills at bedtime on nights 3-10, and 1 pill at bedtime on night 11, then D/C). They return to the Sleep Lab for polysomnography on nights 8 - 10 of medication so their sleep data can be compared.
  Arms: Placebo
Drug: Gabapentin dispensed to subject. — After spending 3 baseline nights in the UM Sleep Lab, alcohol dependent subjects are randomized to receive either gabapentin or placebo for 11 days. (1 pill (600 mg) at bedtime on nights 1 and 2, 2 pills (totalling 1200 mg) at bedtime on nights 3-10, and 1 pill (600 mg) at bedtime on night 11, then D/C). On nights 8 - 10 of medication, subjects return to the lab and sleep 3 more nights with the same procedures.
  Other Names: Neurontin is the brand name for Gabapentin.
  Arms: Gabapentin

SUMMARY:
Insomnia and other sleep abnormalities are common, persistent, and associated with relapse in alcohol-dependent patients. The overall, long-term objectives of the proposed research are to investigate the neurophysiologic mechanisms of sleep disturbance that are associated with relapse in patients with alcohol dependence, and to target those mechanisms with medication in order to reduce relapse risk.

The specific research aims are:

1. To investigate three potential mechanisms of sleep disturbance in alcoholic patients: impaired sleep drive, impaired circadian regulation of alertness, and brain hyperactivation;
2. To investigate short-term effects of medication on sleep and its regulatory mechanisms in alcoholics;
3. To investigate the short-term clinical course of alcoholism as a function of baseline sleep parameters.

In Study Phases I & II (Screening & Baseline: 10+ days), subjects are assessed to diagnose alcohol dependence, determine baseline values for drinking and sleeping, and rule out confounding sleep-impairing causes.

Phase III (Medication: 10 days), is a randomized, double-blind parallel design comparison of gabapentin vs. placebo on mechanisms of sleep. It is not a therapeutic or clinical trial. Phases II & III each have 7 days of monitoring sleep and activity, followed by 3 nights in the University of Michigan (UM) sleep laboratory to assess all-night EEG activity and Dim-Light Melatonin Onset (DLMO), a measure of circadian rhythm.

Phase IV is a 2-day medication taper and Phase V (Follow-up) consists of one visit or telephone call after 12 weeks to assess course of drinking.

In summary, sleep disturbance in alcoholic patients increases their risk of relapse. This study proposes to investigate the mechanisms causing sleep disturbance in alcoholics and to determine if those mechanisms predict return to drinking after 12 weeks.

Relevance: Alcoholism is a devastating chronic disorder that in any one year affects 10% of adults, costs over $185 billion, and causes more than 100,000 deaths in the U.S. Despite treatment, most alcoholic patients achieve only short-term abstinence. Medically-based treatment improvements are needed that target neurophysiologic mechanisms of relapse. Overall public health will be improved by developing science-based treatments that can augment existing, but only partially effective, treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-IV criteria for alcohol dependence (as confirmed by the SCID)
* Between 3 and 12 weeks since last drink (as measured by the TLFB)
* At least 2 weeks since last detoxification medication, if relevant
* An alcohol withdrawal rating score < 8 (as measured by the CIWA-Ar) to rule out acute alcohol withdrawal effects on sleep.
* Expresses a desire to stop drinking or a willingness to abstain from alcohol and/or other drugs of abuse (except nicotine) during the course of the study

Exclusion Criteria:

* Subjects who meet DSM-IV criteria for dependence on any psychoactive substance other than alcohol (except nicotine) in the past 3 months (per SCID interview).
* Subjects with a current (past 1 month) DSM-IV diagnosis of panic disorder, generalized anxiety disorder, post-traumatic stress disorder, major depression, anorexia nervosa, or bulimia nervosa (per SCID interview) and/or that require ongoing psychotropic medication.
* Subjects who have a lifetime diagnosis meeting DSM-IV criteria for bipolar disorder, schizophrenia, schizoaffective disorder, delusional (paranoid) disorders, or obsessive-compulsive disorder.
* Urine drug screen positive for amphetamines, barbiturates, benzodiazepines, cocaine, marijuana, or opioids. (If positive, subjects have one opportunity to test negative after a week of abstinence).
* Medical disorders or pain syndromes that may affect sleep; history of head trauma with loss of consciousness; history of seizures (except alcohol-related seizures).
* Subjects with elevated renal tests (blood urea nitrogen or creatinine), because gabapentin is renally eliminated, or elevated liver transaminases (>3X normal), or abnormal thyroid tests as thyroid problems can affect sleep.
* Sleep disorders other than insomnia such as sleep apnea/hypopnea index >10 per hour or periodic limb movement disorder; PLM>15 movements per hour with arousals.
* Taking medications known to affect sleep (e.g., antidepressants, anticonvulsants, centrally acting antihistamines, neuroleptics, sedative-hypnotics, stimulants, centrally acting antihypertensives [alpha-methyldopa, reserpine, clonidine], oral corticosteroids, and theophylline within the past 2 weeks or 5 weeks for fluoxetine).
* Subjects taking medications used to treat addiction (e.g., disulfiram, naltrexone or acamprosate) are excluded because of unknown effects on sleep.
* Subjects who do evening or midnight shift work. (Subjects who have traveled across multiple time zones in the previous two weeks will be included only at the discretion of the P.I.)
* Pregnancy, breast feeding, or inadequate contraception in women of child-bearing potential.
* Subjects who are unable or unlikely to follow the study protocol in the investigator 's opinion, because of cognitive deficits (Mini-Mental State Exam score < 27), a personality disorder, a serious suicide risk, dangerousness to others, illiteracy, or unstable or distant living situation.
* Subjects with a known allergy, hypersensitivity or contraindication to study medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirk J Brower, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Alcohol-dependent subjects spend 3 nights in the UM sleep lab, then are randomized to receive placebo for one week. They then return to the sleep lab for the same procedures.
  Placebo dispensed to subjects: Alcohol-dependent subjects have polysomnography in the UM Sleep Lab for three nights, then are randomized to receive placebo for 11 days, (1 pill to represent 600mg at bedtime on nights 1 and 2, 2 pills to represent 1200mg at bedtime on nights 3-10, and 1 pill to represent 600mg at bedtime on night 11, then D/C). They return to the Sleep Lab for polysomnography on nights 8 - 10 of medication so their sleep data can be compared.
- Gabapentin: Alcohol-dependent subjects are randomized to receive gabapentin after spending 3 baseline nights in the UM sleep lab. On nights 1 -2 of medication, the dose is 600 mg by mouth 30 min before bedtime. On nights 3-10, the dose is 1200 mg by mouth 30 min before bedtime. On nights 8 -10 of medication, subjects return to the UM sleep lab and complete 3 sleep nights with the same procedures. On night 11, the dose is reduced to 600 mg by mouth 30 min before bedtime, and then stopped.
Period: Overall Study
Arm/Group | Placebo | Gabapentin
Started | 29 | 30
Completed | 24 | 25
Not Completed | 5 | 5
Not completed — Protocol Violation | 3 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — unable to come to appointment | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Alcohol-dependent subjects spend 3 nights in the University of Michigan (UM) sleep lab, then are randomized to receive placebo for one week. They then return to the sleep lab for the same procedures.
  Placebo dispensed to subjects: Alcohol-dependent subjects have polysomnography in the University of Michigan (UM) Sleep Lab for three nights, then are randomized to receive placebo for 11 days, (1 pill to represent 600mg at bedtime on nights 1 and 2, 2 pills to represent 1200mg at bedtime on nights 3-10, and 1 pill to represent 600mg at bedtime on night 11, then D/C). They return to the Sleep Lab for polysomnography on nights 8 - 10 of medication so their sleep data can be compared.
- Gabapentin: Alcohol-dependent subjects are randomized to receive gabapentin after spending 3 baseline nights in the UM sleep lab. On nights 1 and 2 of medication, the dose is 600 mg by mouth 30 min before bedtime. On nights 3-10, the dose is 1200 mg by mouth 30 min before bedtime. On nights 8 -10 of medication, subjects return to the UM sleep lab and complete 3 sleep nights with the same procedures. On night 11, the dose is reduced to 600 mg by mouth 30 min before bedtime, and then stopped.
- Total: Total of all reporting groups
Arm/Group | Placebo | Gabapentin | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (12.5) | 37.0 (8.9) | 36.0 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 23 | 23 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 27 | 26 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 21 | 19 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21 | 19 | 40
  Black | 6 | 7 | 13
  Other | 2 | 4 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 30 | 59

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Total Sleep Time in Stage 2 Sleep Pre- and Post-study Medication (Stage 2 Percent)
Description: Electrophysiological measures of sleep stages: percent of total sleep time in stage 2 sleep
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: percentage of total sleep time
Groups:
- Gabapentin: Alcohol-dependent subjects are randomized to receive gabapentin after spending 3 baseline nights in the UM sleep lab. On nights1 and 2 of medication, the dose is 600 mg by mouth 30 min before bedtime. On nights 3-10, the dose is 1200 mg by mouth 30 min before bedtime. On nights 8 -10 of medication, subjects return to the UM sleep lab and complete 3 sleep nights with the same procedures. On night 11, the dose is reduced to 600 mg by mouth 30 min before bedtime, and then stopped.
Arm/Group | Placebo | Gabapentin
Number analyzed (Participants) | 24 | 25
percentage of total sleep time
  Stage 2 % pre-intervention | 51.3 (8.2) | 53.8 (9.2)
  Stage 2 % post-intervention | 50.2 (7.9) | 59.6 (9.0)

2. Primary Outcome: Wake Time After Sleep Onset (WASO) Measured in Sleep Laboratory Recordings Pre- and Post- Study Medication
Description: Wake time after sleep onset (WASO) (number of minutes awake throughout the night after initial sleep onset)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Gabapentin
Number analyzed (Participants) | 24 | 25
minutes
  pre-intervention | 16.7 (12.5) | 26.5 (19.7)
  post-intervention | 21.9 (20.4) | 14.2 (11.6)

3. Secondary Outcome: Relapse to Any Drinking
Description: Relapse to any drinking is counted as participants who drank any beverage alcohol from end of sleep laboratory study (night 10) to twelve weeks later
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Gabapentin
Number analyzed (Participants) | 24 | 25
Participants | 13 | 14

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | Placebo | Gabapentin
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 2/29 | 4/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=29) | Gabapentin (N=30)
cold (Respiratory, thoracic and mediastinal disorders) | 0 | 2
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
irritability (Psychiatric disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes